CLINICAL TRIAL: NCT03121495
Title: Comparison of Second Forward View Examination and Conventional Withdrawal Examination in the Right Colon on Polyp Detection in Screening and Surveillance Colonoscopies: A Randomized Controlled Study (SFVRC Study)
Brief Title: Study on Second Forward View Examination in the Right Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SFVRC Study
Record Dates: First submitted 2017-04-16; First posted 2017-04-20 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Colonic Polyp; Colorectal Cancer
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Second forward view exam (Active Comparator): During withdrawal, the colonoscope will be advanced to the cecum again when hepatic flexure was reached the first time, where a second forward view (SFV) examination of the right colon will be performed.
  Interventions: Diagnostic Test: Second forward view (SFV) examination of the right colon
- Conventional withdrawal exam (No Intervention): No intervention additional to the conventional withdrawal examination during withdrawal

INTERVENTIONS:
Diagnostic Test: Second forward view (SFV) examination of the right colon — The colonoscope will be advanced to the cecum again when hepatic flexure was reached the first time, where a second forward view (SFV) examination of the right colon will be performed
  Arms: Second forward view exam

SUMMARY:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 2013.

CRC is one of the most preventable cancers because its development in general follows an adenoma-carcinoma sequence. Adenomas are considered precursor lesions for CRC.

While early detection and removal of colorectal adenoma by screening colonoscopy with polypectomy reduce CRC incidence and mortality, interval cancers (cancers that develop after a colonoscopy and before the next scheduled colonoscopy) may still occur and were reported to account for up to 10.5% of CRC. The protective effect of colonoscopy against cancer in the right colon has not been consistently demonstrated. Interval CRC has been associated with proximal colon location, small lesion, flat lesion, missed lesion, inadequate examination, incomplete resection of lesion, tumor biology, and low adenoma detection rate (ADR).

High ADR (eg, ≥ 20%) has been associated with a reduced risk of interval CRC. Methods that can improve polyp detection in the right colon such as retroflexed examination of the right colon, second forward view examination of the right colon, use of colonic fold flattening device, colonoscope with an increased field of view may potentially reduce the risk of interval CRC, but data is still limited. Performance of a second forward view (SFV) examination of the right colon may be the easiest and safest from a practical standpoint when compared to other options (eg, additional training is often needed for retroflexed examination of the right colon since there may be a potentially higher risk of perforation in endoscopists not familiar with the technique, additional equipment is needed when using a colonic fold flattening device, or a colonoscope with an increased field of view).

Our current study aims to determine whether a routine SFV examination in the right colon can lead to an increase in adenoma / polyp detection when compared to conventional withdrawal examination in the right colon in both male and female patients undergoing screening and surveillance colonoscopies.

DETAILED DESCRIPTION:
It is estimated that there are about 1.4 million patients with colorectal cancer (CRC) worldwide, with a rising trend in CRC incidence in many Asian Pacific countries. In Hong Kong, colorectal cancer ranks first in cancer incidence and second in cancer mortality based on data from 2013.

CRC is one of the most preventable cancers because its development in general follows an adenoma-carcinoma sequence. Adenomas are considered precursor lesions for CRC.

While early detection and removal of colorectal adenoma by screening colonoscopy with polypectomy reduce CRC incidence and mortality, interval cancers (cancers that develop after a colonoscopy and before the next scheduled colonoscopy) may still occur and were reported to account for up to 10.5% of CRC. The protective effect of colonoscopy against cancer in the right colon has not been consistently demonstrated. Interval CRC has been associated with proximal colon location, small lesion, flat lesion, missed lesion, inadequate examination, incomplete resection of lesion, tumor biology, and low adenoma detection rate (ADR).

High ADR (eg, ≥ 20%) has been associated with a reduced risk of interval CRC. Methods that can improve polyp detection in the right colon such as retroflexed examination of the right colon, second forward view examination of the right colon, use of colonic fold flattening device, colonoscope with an increased field of view may potentially reduce the risk of interval CRC, but data is still limited. Performance of a second forward view (SFV) examination of the right colon may be the easiest and safest from a practical standpoint when compared to other options (eg, additional training is often needed for retroflexed examination of the right colon since there may be a potentially higher risk of perforation in endoscopists not familiar with the technique, additional equipment is needed when using a colonic fold flattening device, or a colonoscope with an increased field of view).

Our current study aims to determine whether a routine SFV examination in the right colon can lead to an increase in adenoma / polyp detection when compared to conventional withdrawal examination in the right colon in both male and female patients undergoing screening and surveillance colonoscopies.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing colonoscopy for CRC screening or polyp surveillance
* Age 50 - 75 years
* Written informed consent available

Exclusion Criteria

* Contraindications for endoscopy due to comorbidities
* Unable to provide written informed consent
* Personal history of prior resection of any portion of the colon, familial polyposis syndrome, inflammatory bowel disease
* Patients with incomplete colonoscopy (i.e, inability to achieve cecal intubation), a Boston Bowel Preparation Scale (BBPS) score of 0 in either right colon, transverse colon, or left colon at the time of colonoscopy
* Known history of coagulopathy and thrombocytopenia
* Pregnant patients

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1011 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Per-patient ADR in the right colon in each group. | 24 months
  For the SFV group, it is defined as the number of patients with at least 1 adenoma identified in the right colon on either the first or second examination of the right colon divided by the total number of patients in the SFV group. Thus, if a patient has at least 1 adenoma detected on both the first examination and the second examination of the right colon, then this patient will be counted once only. For the conventional group, it is defined as the number of patients with at least 1 adenoma identified in the right colon on the conventional withdrawal examination of the right colon divided by the total number of patients in the conventional withdrawal group.

SECONDARY OUTCOMES:
Increase in per-patient ADR in the right colon in the SFV group. | 24 months
  It is defined as the difference between the new ADR in the right colon after the first examination and SFV (again, if a patient has at least 1 adenoma detected on both the first examination and the second examination of the right colon, then this patient will be counted once only) and the ADR in the right colon after the first examination.
Overall ADR for the entire colon in each group. | 24 months
  For the SFV group, it is defined as the number of patients with at least 1 adenoma identified on either the second examination of the right colon or on the first examination of the right + examination from hepatic flexure to rectum, divided by the total number of patients in the SFV group. Thus, if a patient has at least 1 adenoma detected on both the first examination and the second examination of the right colon, then this patient will be counted once only. For the conventional group, it is defined as the number of patients with at least 1 adenoma identified in the whole colon on the conventional withdrawal examination divided by the total number of patients in the conventional withdrawal group.
The number of patients with at least 1 additional adenoma detected in right colon in the SFV group | 24 months
  For the SFV group, this is the additional adenoma yield on 2nd forward view exam of the right colon
Adverse events during colonoscopy and up to 30 days post colonoscopy | 24 months
  Adverse event rate in SFV group and conventional group
Total number of adenomas found on the first and second examinations of the right colon in the SFV group, and that on the examination of the right colon in the conventional group | 24 months
  This represents the absolute number of adenomas found on the first and second examinations of the right colon in the SFV group, and that on the examination of the right colon in the conventional group
Total number of polyps found on the first and second examinations of the right colon in the SFV group, and that on the examination of the right colon in the conventional group | 24 months
  This represents the absolute number of polyps found on the first and second examinations of the right colon in the SFV group, and that on the examination of the right colon in the conventional group

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tang, MD, Principal Investigator — Institute of Digestive Disease, The Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang RSY, Lee JWJ, Chang LC, Ong DEH, Chiu HM, Matsuda T, Kim HS, Sekiguchi M, Leong RW, Ho AMY, Lam TYT, Tse YK, Lin L, Yeoh KG, Lau JYW, Sung JJY; Asia Pacific Working Group on Colorectal Cancer Screening. Two vs One Forward View Examination of Right Colon on Adenoma Detection: An International Multicenter Randomized Trial. Clin Gastroenterol Hepatol. 2022 Feb;20(2):372-380.e2. doi: 10.1016/j.cgh.2020.10.014. Epub 2020 Oct 14. PMID 33065307

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03121495/Prot_SAP_000.pdf